CLINICAL TRIAL: NCT03746678
Title: Patient-Centered Perioperative Care Through Mobile Application: Patient Engagement Prospective Cohort Study in Elective Cesarean Delivery Patients
Brief Title: Patient-Centred Perioperative Mobile Application
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IWK Health Centre (Other)
Responsible Party: Sponsor
Other Study IDs: IWK1023201
Record Dates: First submitted 2018-11-05; First posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Cesarean Delivery
Keywords: Cesarean delivery; Perioperative medicine; Mobile health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- C-Care Mobile Application
  Interventions: Other: C-Care Mobile Application

INTERVENTIONS:
Other: C-Care Mobile Application — C-care is a mobile application developed based on previous research at the IWK Health Centre. It contains topics relevant to Cesarean delivery and the recovery process, which the patient could access at anytime. Patient engagement with the application will be monitored anonymously for 30 days after delivery. On days one to five after delivery, patients will receive a short self-monitoring questionnaire (approximately 1 minute). At the end of two weeks (14 days), patients will complete an online survey regarding overall satisfaction, potential impact on care, usability and feasibility problems. At any point during the study, patients can email us to report any problems with the application.

SUMMARY:
With increasingly more complex surgical patients and the trend toward decreased hospital stay after operations, continuity of care and prompt management of symptoms and side effects perioperatively are ever more crucial. The investigators' goal is to improve perioperative care with a patient-centred mobile application, starting with a pilot in patients undergoing elective Cesarean delivery. The investigators have completed a research study where they created a prototype based on feedback from patients and anesthesiologists. In this study, the investigators would like to learn about how patients use our mobile application after delivery and how the mobile application can be integrated into daily practice.

DETAILED DESCRIPTION:
The objective of this cohort study is to build the mobile application and evaluate its feasibility in providing patient education and reminders for self-monitoring for cesarean delivery patients. The investigators will measure the extent of patient engagement with our application through in-app usage data, as well as receive quantitative and qualitative feedback regarding feasibility. By understanding user behavior and needs through questionnaires and application usage data, the investigators could design more effective and tailored interventions for patients. Results of this study will help further development and implementation of an interdisciplinary mobile monitoring and communication platform for perioperative care.

This study is funded by the Dalhousie University Department of Anesthesia, Pain Management & Perioperative Medicine.

ELIGIBILITY:
Inclusion Criteria:

Part 1 (screened by asking nurse)

* Patient scheduled for elective Cesarean delivery
* Age equal or greater than 18
* American Society of Anesthesiologists (ASA) Physical Status I-III (i.e. not in life-threatening situation)

Part 2 (screened in person)

* Possesses an iOS Smartphone with active data plan and access to WiFi, and self-reported use of it on a regular basis (at this stage in development, the mobile application prototype is only available on iOS)
* Self-reported proficiency with Smartphone and mobile applications
* Reported fluency in English

Exclusion Criteria:

Self-reported physical or psychiatric condition that may impair the ability to use the mobile application, answer questionnaires and surveys, and/or provide insights representative of the general population, such as blindness, under current influence of recreational drugs or alcohol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective Cesarean delivery patients at the IWK Health Centre
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2018-11-19 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Median number of information topics viewed per participant | 30 days
  Quantitative mobile application usage data
Median number of self-monitoring questionnaires completed per participant | 30 days
  Quantitative mobile application usage data
Median number of total visits to the mobile application per participant | 30 days
  Quantitative mobile application usage data
Satisfaction score (scale of 0 to 10, 10 being extremely satisfied, 0 being not satisfied) | 2 to 3 weeks
  Quantitative responses from survey
Percentage of participants who would recommend the C-Care App to other women undergoing Cesarean delivery | 2 to 3 weeks
  Quantitative responses from survey
Percentage of self-monitoring questionnaires completed (out of 5) per participant | 30 days
  Quantitative mobile application usage data

SECONDARY OUTCOMES:
Which topics were viewed the most (rank by topic name and by postoperative day) | 30 days
  Quantitative mobile application usage data
Which self-monitoring questionnaires were filled the most (rank by postoperative day number) | 30 days
  Quantitative mobile application usage data
Incidence of important potential anesthetic-related problems entered by the patient (pain, headache, weakness and numbness) | 30 days
  Quantitative mobile application usage data
Time of the day patient visited site (scatter plot of Nova Scotia time vs. # visits) - one visit = at least one interaction within app, e.g. opening a topic, navigating within app | 30 days
  Quantitative mobile application usage data
Time of the day patient filled out the questionnaire | 30 days
  Quantitative mobile application usage data
Number of visits vs. postoperative day | 30 days
  Quantitative mobile application usage data
Median duration (number of days starting from delivery date until the last day of visit) patient interacted with application. | 30 days
  Quantitative mobile application usage data
% participant who responded "yes" to the question that C-Care App provided them with knowledge about Cesarean delivery and anesthesia | 2 to 3 weeks
  Quantitative responses from survey
% participant who responded "yes" to the question that C-Care App provided them with knowledge about potential complications to monitor for | 2 to 3 weeks
  Quantitative responses from survey
% participant who responded "yes" to the question that C-Care App provided them with knowledge about the recovery process after Cesarean delivery | 2 to 3 weeks
  Quantitative responses from survey
Anything the patient wanted to change about this application, in terms of content, navigation, appearance, and overall experience? | 2 to 3 weeks
  Qualitative responses from survey
If the patient did not use the mobile application, what were the reasons? | 2 to 3 weeks
  Qualitative responses from survey
How could we make the mobile application more helpful for the patient? | 2 to 3 weeks
  Qualitative responses from survey
What do patients think about the name of this App, "C-Care"? Do they have any other suggestions for our name/logo? | 2 to 3 weeks
  Qualitative responses from survey
Any other comments and/or suggestions | 2 to 3 weeks
  Qualitative responses from survey

CONTACTS AND LOCATIONS:
Locations (1):
- Women's and Obstetric Anesthesia, IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ke JXC, George RB, Wozney L, Munro A. Perioperative mobile application for mothers undergoing Cesarean delivery: a prospective cohort study on patient engagement. Can J Anaesth. 2021 Apr;68(4):505-513. doi: 10.1007/s12630-020-01907-x. Epub 2021 Jan 9. PMID 33420678
- See also: C-Care mobile application prototype — https://itunes.apple.com/ca/app/c-care/id1373322196?mt=8

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT03746678/Prot_SAP_000.pdf